CLINICAL TRIAL: NCT03225768
Title: Adopting Guided Training to Improve Participation Performance of Individuals With Cognitive Impairments After Stroke and Traumatic Brain Injury: A Feasibility Study (GTPCI)
Brief Title: Guided Training for People With Cognitive Impairment
Acronym: GTPCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yen-Nung Lin, Director of Rehabilitation Department of Taipei Medical University WanFang Hospital, Taipei Medical University WanFang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N201704046
Record Dates: First submitted 2017-06-22; First posted 2017-07-21 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: TBI (Traumatic Brain Injury); Stroke; Cognitive Impairment
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke; Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guided Training (Experimental)
  Interventions: Behavioral: Guided Training

INTERVENTIONS:
Behavioral: Guided Training — Guided training is an intervention strategy designed to help individuals identify barriers in their daily life and guide them to generate their own strategies to address these barriers. This intervention strategy is different from traditional direct skill training, in which rehabilitation practitioners are responsible for identifying their patients' challenges to perform activities and teaching them task-specific problem-solving strategies. Guided training has been applied in a variety of clinical populations, including individuals with stroke and TBI, and has demonstrated significant effect on improving independence with daily activities among persons with acute stroke-related cognitive impairments enrolled in inpatient rehabilitation.

SUMMARY:
Abstract

Objective: Investigators examined the feasibility of applying a participation-focused strategy training intervention to community-dwelling adults with cognitive impairments following stroke and brain injury and evaluated its potential effect on participation.

Method: Participants with a diagnosis of stroke or brain injury participated in this single-group, repeated-measures study. Participants received 1~2 sessions of strategy training intervention weekly for 8~18 sessions. Outcome measures included the Participation Measure--3 Domains, 4 Dimensions (PM-3D4D), the Canadian Occupational Performance Measure (COPM), and feasibility indicators (participants' recruitment, retention, attendance, engagement, comprehension, satisfaction, and intervention adherence).

DETAILED DESCRIPTION:
Method

Design A single-group, repeated-measures design was adopted for this study. All participants received the participation-focused strategy training intervention and the assessments at baseline (T1) and at post-intervention (T2). The study protocols were approved by the university institutional review board.

Intervention

The intervention protocols were developed based on the strategy training guidelines developed by Skidmore et al. Three trained research occupational therapists delivered the intervention to participants in addition to their regular outpatient rehabilitation care. The following standardized procedures were followed. First, the therapists asked the participants to identify three participation goals that they perceived important to them. Next, the participants were asked to identify barriers to their performance, and according to which the therapists taught the participants the "Goal-Plan-Do-Check" strategy, which involves (1) setting a goal to address the barriers, (2) developing a plan to address the goal, (3) doing the plan, and (4) checking if the plan worked or required revising. This procedure repeated iteratively until the participants' goal was met, and the next goal could be moved on to. At the end of each session, the therapists prompted the participants to identify the principles they learned during the session and encouraged the participants to apply these principles in the next session. Each participant received 1~2 intervention sessions per week for a total of 10~20 intervention sessions (or until their goals were achieved) from trained research therapists. Each session lasted for 45~60 minutes. All intervention sessions were recorded and rated for fidelity by research staff.

Measures

Background Characteristics. Demographic variables (e.g., age and gender) were collected through a questionnaire developed by the research team at baseline assessment. Clinical variables (e.g., diagnosis and time since injury/illness) were retrieved from participants' medical charts.

Feasibility Indicators. Investigators assessed feasibility by examining (1) the number of participants recruited and retained; (2) the number of intervention sessions that participants attended; (3) participants' engagement in the intervention sessions (assessed by the research therapists using the Pittsburgh Rehabilitation Participation Scale, measured on a 6-point scale: 1: no engagement to 6: excellent engagement); (4) participants' comprehension of the intervention sessions (assessed by a 3-point scale: 1: minimal understanding to 3: good understanding); (5) participants' satisfaction with the intervention (assessed by the Client Satisfaction Questionnaire, a 8-item questionnaire, with total scores 8~32 (0~23: poor to fair satisfaction; 24~32: moderate to high satisfaction); and (6) the intervention adherence (measured by the Strategy Training Fidelity Checklist, for which an independent rater randomly selected 20% of sessions to rate the research therapists' adherence to the principles in the intervention protocol (yes, no) and competence in execution (inadequate, adequate, exceptional).

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria include that the participant:

1. ages 20 years and older;
2. had a first-time stroke or TBI;
3. is able to understand Mandarin;
4. has cognitive impairment (indicated by a score of 25 or less on the Montreal Cognitive Assessment (MoCA) or a score of 3 or less on the executive function subsection of MOCA);
5. is able to provide informed consent.

Exclusion Criteria:

Participants will be excluded if they:

1. have severe aphasia
2. have a pre-stroke diagnosis of dementia, current major depression disorder, substance use, or other psychiatric disorders that may impede them from continually participating in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-11-18 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | From baseline to 6 months following the completion of the intervention
  The PM-3D4D is a 19-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community, rated on four dimensions: (1) 'Diversity of participation' (yes [1] vs. no [0]); (2) 'Frequency' (5- and 7-point scales, from "never" to "everyday or almost everyday"); (3) 'Desire for change' (yes [1] vs. no [0]); and (4) 'Perceived difficulty' (4-point scale, from "very difficult" [1] to "not difficult at all" [4]). Each dimensional score of the PM-3D4D can be separately summed for each domain. Psychometric properties of the PM-3D4D were established in rehabilitation populations.
Canadian Occupational Performance Measure (COPM) | From the first session to the last session of the intervention, up to 10 weeks
  The COPM inquires the client to identify important goals in their daily life and rate their performance and satisfaction for each goal on a 10-point visual analog scale.

SECONDARY OUTCOMES:
Activities | From baseline to 6 months following the completion of the intervention
  Activity Measure for Post-Acute Care (AM-PAC) Outpatient Short Forms
Cognitive functioning | From baseline to 6 months following the completion of the intervention
  Wisconsin Card Sorting Task (WCST)

CONTACTS AND LOCATIONS:
Locations (1):
- WanFang Hospital, New Taipei City, Taiwan